CLINICAL TRIAL: NCT03862898
Title: Efficacy of the Lumbar Stabilization and Thoracic Mobilization Exercise Program on Pain Intensity and Functional Disability Reduction in Chronic Low Back Pain Patients: a Randomized Controlled Single-blind Trial
Brief Title: Efficacy of the Lumbar Stabilization and Thoracic Mobilization Exercises in Chronic Low Back Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stefan Kostadinović (Other)
Responsible Party: Sponsor-Investigator, Stefan Kostadinović, Principal Investigator, University of Novi Sad
Organization: University of Novi Sad (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01-39/122/1
Record Dates: First submitted 2019-03-02; First posted 2019-03-05 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lumbar stabilization group- thoracic (Experimental): Lumbar stabilization and thoracic mobilization in a closed kinetic chain (LSTMC) group performed this exercises from the least to the largest painless motion amplitude and accordingly divided into three phases. The first phase lasted for two weeks, the second three and the last third phase, also for three weeks, and a total of 8 weeks.
  Interventions: Other: Lumbar stabilization exercises
- lumbar stabilization group (Active Comparator): Lumbar stabilization in a closed and opened kinetic chain (LSCO) group also performed exercises from the least to the largest painless motion amplitude in three phases.
  Interventions: Other: Lumbar stabilization exercises

INTERVENTIONS:
Other: Lumbar stabilization exercises — Patients performed exercises to stabilize and strengthen paravertebral muscles. Three sets of ten repetitions with a minute break between each.

SUMMARY:
Chronic low-back pain (CLBP) is a heterogeneous group of disorders, which according to the new classification of the International Association for Pain Research (IASP), is recognized as an independent entity and belongs to a mixed type of pain caused by central sensitization , which is present for more than 12 weeks. Studies have found that lumbar segmental instability (LSI) is one of the most significant cause of lumbar pain through the movement of each spinal segment where degenerative changes were observed in the discs. The aim of this study was to compare the program of lumbar stabilization exercises in the open and closed kinetic chain, in relation to the program of lumbar stabilization exercises and thoracic mobilization in a closed kinetic chain, to evaluate the clinical efficacy of both exercise programs and determine whether initial pain intensity values and disability levels affect the outcome of patients with chronic low back pain. The study was conducted as randomized, single-blind, controlled trial in 80 chronic low-back pain (CLBP) patients of both sexes (35 male, 45 female), average age (48.45 +/- 10.22 years, treated at the Rehabilitation Clinic "Dr. Miroslav Zotović" in Belgrade between June 2017 and March 2018. Respondents were divided into two groups of 40 patients by simple randomization. Participants were given laser therapy, transcutaneous electrical nerve stimulation (TENS) and an eight-week kinesiotherapy that included exercises to strengthen the deep lumbar spine stabilizers. Retesting was done after 4 and 8 weeks. Patients who performed lumbar stabilization and thoracic mobilization exercises program in a closed kinetic chain had better functional recovery and a significant reduction in pain intensity compared to respondents who performed a lumbar stabilization program in opened and closed kinetic chain.

ELIGIBILITY:
Inclusion Criteria:

* patients with lumbar pain present for more than 12 weeks,
* pain during changing of the position,
* radicular pain.

Exclusion Criteria:

* Cauda equina syndrome,
* ankylosing spondylitis,
* thoracic deformities (pectus carinatum, excavatum),
* spina bifida,
* fractures,
* post-operative spinal conditions,
* diabetes,
* inflammatory processes,
* tumors,
* pregnancy.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Pain intensity | eight weeks
  According to Visual Analogue scale, pain intensity was assessed for lumbosacral spine and for the leg in mm. On the graphic scale, there is a horizontal line of 10 cm. The beginning of the line with 0 is marked, which indicates that there is no pain, the middle with 5 and the end with 10, which marks the strongest pain. The respondents are asked to mark the site, which most closely indicates the intensity of his pain in the back in the past 24 hours, and then on the scale mark the severity of pain in the back and legs. After that, the ruler measures the obtained value in the millimeters and they are entered
Functional disability | eight weeks
  According to Oswestry disability Index, functional disability was assessed. This index contains ten categories of six questions. The intensity of pain, the ability to raise loads, take care of oneself, walk, sit, sexual functions, standing, social life, the quality of sleep and traveling. The patient completes the label in front of him, which most resembles his situation. Each category is scored on a scale of 0-5, where the first statement is zero and indicates the smallest amount of incapacity, and the last statement of 5 points shows a very difficult degree of disability.

SECONDARY OUTCOMES:
Dolour Neuropathic test (DN4) | eight weeks
  It is a questionnaire for assessing the neuropathic component of pain. Consists of four questions. Answers to the first two are obtained on the basis of an interview with the patient and they speak of the character of the pain, and the other two, based on a clinical examination. In the first, three responses are offered, in the second four, the third two, and in the last question, one answer. The respondent does not have to give an answer, and can respond to more than one offered. If the patient's score is 4 or greater, the test indicates that there is a specificity greater than 90% for the test subjects in determining the neuropathic pain component
Prone instability test | eight weeks
  This test is performed by exposing the spinosus process of the lumbar spine to the hypothenar, while the patient is in the stomach position at the edge of the table, with toes on the floor. When the subject reports pain, the examiner instructs him to lift his fingers from the floor and lift his legs to a horizontal position. If the patient now has no discomfort or pain, the test is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Ljubica Konstantinovic, Phd, Study Chair — Clinic for rehabilitation "dr Miroslav Zotović", Belgrade
Locations (1):
- Clinic for rehabilitation "dr Miroslav Zotović", Belgrade, Serbia